CLINICAL TRIAL: NCT00117468
Title: A Phase 2, Single-Center, Open-Label, Randomized, Controlled, Pharmacodynamic Study to Compare DR-2011 to a Progesterone Vaginal Gel for Luteal Phase Replacement
Brief Title: Comparison of DR-2011 to a Progesterone Vaginal Gel for Luteal Phase Replacement
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duramed Research (Industry)
Responsible Party: Duramed Protocol Chair, Duramed Research, Inc.
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DR-PGN-201
Record Dates: First submitted 2005-06-30; First posted 2005-07-07 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-05

CONDITIONS: Infertility
Keywords: luteal phase replacement; oocyte donation; infertility; progesterone
MeSH Terms: conditions — Infertility | interventions — Progesterone; Vaginal Creams, Foams, and Jellies; Crinone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: DR-2011
- 2 (Active Comparator)
  Interventions: Drug: Progesterone 8% Vaginal Gel

INTERVENTIONS:
Drug: DR-2011 — Administered vaginally from Day 14 to Day 31
  Arms: 1
Drug: Progesterone 8% Vaginal Gel — Administered vaginally from Cycle Day 14 to Day 31
  Other Names: Crinone
  Arms: 2

SUMMARY:
This is a single-center, open-label, randomized, active-controlled study to compare DR-2011 to progesterone vaginal gel for luteal phase replacement.

DETAILED DESCRIPTION:
This is a 2-arm, single-center, open-label, randomized, active-controlled study to compare the safety and efficacy of luteal phase replacement with DR-2011 to progesterone vaginal gel over an 18-day treatment period. Patients will also be required to use an estrogen patch during the course of the study. The overall study duration for each patient will be approximately 1½ months.

Luteal phase replacement will be monitored by endometrial biopsy on Cycle Day 25 or 26. In addition, serum hormonal levels will be measured at screening and at designated times from Cycle Day 14 to 31.

ELIGIBILITY:
Inclusion Criteria:

* Not pregnant
* Clinically or medically-induced non-functioning or surgically removed ovaries
* Clinical investigator believes patient would be eligible for oocyte donation

Exclusion Criteria:

* Any contraindication to progesterone or estrogen therapy
* Undiagnosed vaginal bleeding
* History of uterine fibroids or any other conditions that could adversely affect pregnancy success
* Hysterectomy
* Any contraindication to vaginal drug delivery systems

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2005-06; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Adequate endometrial transformation | Cycle Day 25 or 26

SECONDARY OUTCOMES:
Hormone levels | Duration of study

CONTACTS AND LOCATIONS:
Overall Officials: Duramed Protocol Chair, Study Chair — Duramed Research, Inc,
Locations (1):
- Duramed Investigational Site, Norfolk, Virginia, United States

REFERENCES:
- See also: MedlinePlus - Infertility — http://www.nlm.nih.gov/medlineplus/infertility.html